CLINICAL TRIAL: NCT00106223
Title: A Randomized Waitlist Controlled Treatment Trial Investigating CBT for Body Dysmorphic Disorder
Brief Title: Treatment Study Investigating New Cognitive Behavioral Therapy Treatment Manual for Body Dysmorphic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sabine Wilhelm, PhD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH070490 (NIH); R34MH070490 (NIH); 2004-P-000478/7; DATR A2-AIR
Record Dates: First submitted 2005-03-21; First posted 2005-03-22 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Body Dysmorphic Disorder; Somatoform Disorders
Keywords: Cognitive Behavioral Therapy; CBT; BDD; Body dysmorphic disorder
MeSH Terms: conditions — Body Dysmorphic Disorders; Somatoform Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Group receiving immediate treatment with cognitive behavioral therapy
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)
- 2 (Active Comparator): Waitlist control group to begin CBT 3 months after other CBT group begins treatment
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) — Participants will receive a total of 22 sessions of individual, manual-based CBT. The CBT sessions will occur weekly during the course of the study. During the sessions, participants will receive education about BDD and CBT, engage in activities that help them confront their BDD, learn new ways of thinking about body image, and learn relapse prevention techniques.
  Other Names: CBT

SUMMARY:
In an earlier phase of this study, a cognitive behavioral therapy (CBT) manual to treat body dysmorphic disorder (BDD) symptoms was developed. We are currently implementing this manual-based treatment to validate its effectiveness in patients with BDD.

DETAILED DESCRIPTION:
BDD is a disease that involves preoccupation with imagined or minor physical flaws. The condition often begins in adolescence and, if left untreated, can cause significant social, emotional, and occupational distress. Within the last decade, BDD has received increased attention, and various modes of treatment have been utilized and evaluated. CBT has been found to be a more effective form of treatment than other types of psychotherapy. In this study, we have created a new CBT treatment manual and are currently implementing it to evaluate its effectiveness in patients with BDD. The utility of this manual for different populations will also be evaluated, and adherence and competence measures to assess CBT delivery will be developed.

This study will last 24 weeks. Participants will be randomly assigned (like the flip of a coin) to either start CBT treatment immediately or to a waitlist group, which would require a 3-month wait without treatment before beginning treatment for this study. Participants have a 50-50 chance of being in either group. Participants will receive a total of 22 sessions of individual, manual-based CBT. The CBT sessions will occur weekly during the course of the study. During the sessions, participants will receive education about BDD and CBT, engage in activities that help them confront their BDD, learn new ways of thinking about body image, and learn relapse prevention techniques. Self-report scales will be used to assess participants.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of BDD for at least 6 months prior to study entry
* Score higher than 23 on BDD Yale-Brown Obsessive Compulsive Scale
* Live within driving distance of Boston, MA or Providence, RI

Exclusion Criteria:

* Any psychiatric diagnoses other than BDD
* Alcohol abuse or dependence within 3 months prior to study entry
* Suicidal or homicidal
* Psychotropic medication within 2 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Body dysmorphic disorder symptoms | Measured at Months 6 and 9

SECONDARY OUTCOMES:
Functioning and life satisfaction | Measured at Months 6 and 9
Depressive symptoms | Measured at Months 6 and 9
Anxiety symptoms | Measured at Months 6 and 9

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, PhD, Principal Investigator — BDD Clinic Director, Massachusetts General Hospital
Locations (2):
- United States (2):
  - BDD Clinic, Massachusetts General Hospital, Charlestown, Massachusetts
  - Body Image Program, Butler Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Fang A, Steketee G, Keshaviah A, Didie E, Phillips KA, Wilhelm S. Mechanisms of Change in Cognitive Behavioral Therapy for Body Dysmorphic Disorder. Cognit Ther Res. 2020 Jun;44(3):596-610. doi: 10.1007/s10608-020-10080-w. Epub 2020 Feb 4. PMID 38031584
- See also: Click here for information on the Body Dysmorphic Disorder Clinic, Massachusetts General Hospital Web site — http://www.massgeneral.org/bdd